CLINICAL TRIAL: NCT03547427
Title: Enhancement of Glucagon Counterregulation in Type 1 Diabetes by Basal Amylin Replacement
Brief Title: Glucagon Counterregulation in Type 1 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical staffing issues and COVID-19 pandemic
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Leon Farhi, PhD, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20364
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Pramlintide; Lispro Insulin; Continuous Glucose Monitor (CGM); Acetaminophen; Hypoglycemia; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Insulin hypoglycemia + pramlintide (Experimental): Subjects will have a 25% reduction in their standard basal insulin therapy with concurrent basal pramlintide infusion ('Basal pramlintide and reduced basal insulin'). They will receive a Lispro bolus to induce hypoglycemia of ≤55mg/dL ('Insulin-induced hypoglycemia'). After induction of hypoglycemia is completed subjects will have an acetaminophen test. Subjects will be instructed to initiate a CGM session 2-3 days prior to both the admissions. Blood samples will be collected during the hypoglycemic induction and acetaminophen test.
  Interventions: Other: Basal pramlintide and reduced basal insulin; Other: CGM; Other: Acetaminophen test; Other: Insulin-induced hypoglycemia
- Insulin hypoglycemia (Active Comparator): Subjects will have their standard basal insulin treatment ('Basal insulin alone') and receive a Lispro bolus to induce hypoglycemia of ≤55mg/dL ('Insulin-induced hypoglycemia'). After induction of hypoglycemia is completed subjects will have an acetaminophen test. Subjects will be instructed to initiate a CGM session 2-3 days prior to both the admissions. Blood samples will be collected during the hypoglycemic induction and acetaminophen test.
  Interventions: Other: Basal insulin alone; Other: CGM; Other: Acetaminophen test; Other: Insulin-induced hypoglycemia
- Exercise hypoglycemia + pramlintide (Experimental): Subjects will have a 25% reduction in their standard basal insulin therapy with concurrent basal pramlintide infusion ('Basal pramlintide and reduced basal insulin'). They will have three bouts of exercise to induce hypoglycemia of ≤55mg/dL ('Exercise-induced hypoglycemia'). After induction of hypoglycemia is completed subjects will have an acetaminophen test. Subjects will be instructed to initiate a CGM session 2-3 days prior to both the admissions. Blood samples will be collected during the hypoglycemic induction and acetaminophen test.
  Interventions: Other: Basal pramlintide and reduced basal insulin; Other: CGM; Other: Acetaminophen test; Other: Exercise-induced hypoglycemia
- Exercise hypoglycemia (Active Comparator): Subjects will have their standard basal insulin treatment ('Basal insulin alone'). They will have three bouts of exercise to induce hypoglycemia of ≤55mg/dL ('Exercise-induced hypoglycemia' ). After induction of hypoglycemia is completed subjects will have an acetaminophen test. Subjects will be instructed to initiate a CGM session 2-3 days prior to both the admissions. Blood samples will be collected during the hypoglycemic induction and acetaminophen test.
  Interventions: Other: Basal insulin alone; Other: CGM; Other: Acetaminophen test; Other: Exercise-induced hypoglycemia

INTERVENTIONS:
Other: Basal insulin alone — A study insulin pump containing lispro insulin will be programmed to deliver basal lispro insulin at according to the subject's normal basal profile. The carbohydrate ratio(s) and insulin sensitivity factor(s) will be programmed per the subject's usual home parameters.
  Arms: Exercise hypoglycemia; Insulin hypoglycemia
Other: Basal pramlintide and reduced basal insulin — A study insulin pump containing pramlintide will be programmed to deliver pramlintide at 6:1 pramlintide:insulin ratio. Simultaneously, a study insulin pump containing lispro insulin will be programmed to deliver basal lispro insulin at ~25% reduced rate from the subject's normal basal profile. The carbohydrate ratio(s) and insulin sensitivity factor(s) will be programmed per the subject's usual home parameters.
  Arms: Exercise hypoglycemia + pramlintide; Insulin hypoglycemia + pramlintide
Other: CGM — Subjects will be instructed to initiate a Continuous Glucose Monitor (CGM) session 2-3 days prior to both the experimental and control CRU admissions.
Other: Acetaminophen test — Consumption of a standardized meal mixed with added 1.5 g liquid acetaminophen
Other: Insulin-induced hypoglycemia — During insulin-induced hypoglycemia admission, subjects will receive an insulin bolus(s) dosed to reach blood sugar of less than 55 mg/dL.
  Arms: Insulin hypoglycemia; Insulin hypoglycemia + pramlintide
Other: Exercise-induced hypoglycemia — During exercise-induced hypoglycemia admission, subjects participate in three 15 minute exercise bouts (45 minutes total) to lower blood sugar to less than 55 mg/dL.
  Arms: Exercise hypoglycemia; Exercise hypoglycemia + pramlintide

SUMMARY:
The purpose of this study is to find out whether the combination of insulin and pramlintide is better than insulin alone at helping the pancreas release glucagon in response to a low blood sugar episode.

A secondary goal is to assess whether basal pramlintide will delay gastric emptying.

DETAILED DESCRIPTION:
Participation in this study will require three (3) study visits over 12 weeks: one screening visit lasting 2-3 hours, and two overnight study visits at the university's Clinical Research Unit (CRU). The two overnight visits will last about 22 hours.

During the CRU admission, all subjects will wear a Continuous Glucose Monitor (CGM) starting 2-3 days prior to the CRU admission and after having a CGM training.

Eligible subjects will be randomized to either insulin- or exercise-induced hypoglycemia group. Each subject will have two overnight CRU admissions in randomized order: Experimental (basal pramlintide + 25% reduction of basal insulin) or Control (standard basal insulin therapy) admissions. During these two admissions, the study team will deliberately induce hypoglycemia as follows:

Subjects randomized to insulin-induced hypoglycemia admission will receive an insulin bolus(s) dosed to reach blood sugar of less than 55 mg/dL.

Subjects randomized to exercise-induced hypoglycemia will participate in three 15 minute exercise bouts (45 minutes total) to lower blood sugar to less than 55 mg/dL.

After hypoglycemia induction, all subjects will receive one and the same standard meal (lunch) mixed with 1.5 g liquid acetaminophen to measure how quickly acetaminophen is absorbed to estimate the rate of gastric emptying.

The study team will collect blood samples during the hypoglycemic induction and the gastric emptying monitoring which will be analysed for levels of various substances used to address the study goals.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least 5 years and using insulin for at least 5 years
* Use of an insulin pump for at least 6 months with established parameters for basal rate(s), carbohydrate ratio(s) and insulin sensitivity factor(s) for at least 3 months.
* HbA1c level <10.5% at screening
* Demonstration of proper mental status and cognition for the study
* Investigator has confidence that the subject can successfully operate all study devices and is capable of adhering to the protocol

Exclusion Criteria:

* Admission for diabetic ketoacidosis in the 6 months prior to enrollment.
* Severe hypoglycemia resulting in seizure or loss of consciousness in the 3 months prior to enrollment.
* Hematocrit less that the lower limit of normal for the assay.
* Pregnancy, breast-feeding, or intention of becoming pregnant over time of study procedures
* A known medical condition, which in the opinion of the investigator or designee, would put the participant or study at risk
* A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol
* Current use of some drugs and supplements
* Participation in another pharmaceutical or device trial at the time of enrollment or during the study
* Basal insulin rates less than 0.01 units per hour
* Diagnosed food allergies that would prohibit the consumption of a standardized meal
* Any reason the study MD considers that the subject is not appropriate for the trial

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Relative glucagon counterregulation (GCR) response | about 19 hours
  The primary outcome is the relative glucagon counterregulation (GCR) response, computed as the ratio between average glucagon concentration in response to insulin-induced hypoglycemia, and the pre-hypoglycemic baseline value. The baseline glucagon level is defined as the average concentration of glucagon when the falling plasma glucose is below 100mg/dl but above the hypoglycemic threshold of 60mg/dl. The response to hypoglycemia is the average concentration of glucagon between the hypoglycemic threshold crossing point and the time of the meal ingestion.

SECONDARY OUTCOMES:
Maximal glucagon counterregulation (GCR) response | about 19 hours
  The maximal glucagon concentration achieved during the response to hypoglycemia
Rate of gastric emptying | about 4 hours
  The time to reaching ½ maximal acetaminophen concentration in the bloodstream after ingesting a meal mixed with 1.5 g of liquid acetaminophen.

CONTACTS AND LOCATIONS:
Overall Officials: Leon S. Farhy, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
To be determined
Time Frame: To be determined
Access Criteria: To be determined